CLINICAL TRIAL: NCT06295523
Title: Heat Waves and the Elderly With COPD: Reducing Thermal and Cardiovascular Consequences
Brief Title: Heat Waves and the Elderly With COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to recruitment challenges coupled with our focus changing to a different direction.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Craig Crandall, Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STU_2019_1759_COPD
Record Dates: First submitted 2024-02-26; First posted 2024-03-06 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: COPD; Aging; Hyperthermia
Keywords: COPD; heat wave; thermoregulation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Very hot and dry (Experimental): Subjects will be exposed to 3 hours in a climate chamber set to approximately 47 deg C and 15% relative humidity, which reflects a very hot and dry heat wave condition similar to the 2018 Los Angeles heat wave. Two visits will be required to complete this arm, with one visit including water spray for cooling.
  Interventions: Other: Water Spray; Other: Control
- Experimental: Hot and humid (Experimental): Subjects will be exposed to 3 hours in a climate chamber set to approximately 41 deg C and 40% relative humidity, which reflects hot and humid heat wave similar to the 1995 Chicago heat wave. Two visits will be required to complete this arm, with one visit including water spray for cooling.
  Interventions: Other: Water Spray; Other: Control

INTERVENTIONS:
Other: Water Spray — Participants will receive water spraying on their body throughout the climate chamber exposure.
Other: Control — Participants will NOT receive water spraying on their body throughout the climate exposure.

SUMMARY:
The purpose of this study is to investigate thermoregulatory responses in older individuals with COPD.

DETAILED DESCRIPTION:
Heat waves are the leading cause of death among natural disasters in the United States.

Elderly individuals are disproportionately more likely to become ill or die during heat waves. While the elderly have a reduced ability to regulate their body temperature,8-10 hospitalizations and deaths in this population during heat waves are primarily due to cardiovascular and/or respiratory complications, not solely hyperthermia. While previous research has primarily focused on the thermal and cardiovascular consequences of healthy aging, very little research has focused on the physiological responses to heat exposure in older individuals with chronic disease, such as chronic obstructive pulmonary disease (COPD). Notably, epidemiological data suggests that pulmonary complications are a leading cause of heat wave-related hospitalizations in older adults with a diagnosis of COPD, yet nothing is known regarding the physiological mechanisms by which those with COPD are most susceptible to heat waves. To fill this important gap, the investigators will identify the physiological responses that occur in this population, relative to healthy age-matched individuals, during two unique heat wave simulations.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or older
* Diagnosis of COPD

Exclusion Criteria:

* Known heart disease
* Other chronic medical conditions requiring regular medical therapy including cancer, diabetes, uncontrolled hypertension, and uncontrolled hypercholesterolemia etc
* Abnormality detected on routine screening suggestive of provokable ischemia or previously undetected cardiac disease or resting left bundle branch block on screening electrocardiogram
* Current smokers
* Participant with a body mass index ≥31 kg/m2

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Core body temperature | Prior to and throughout each simulated heat wave exposure, an average of 480 minutes
  Core body temperature will be measure from gastrointestinal temperature via an ingestible telemetric pill
Forced expiratory volume (FEV1) | Prior to, during, and after each simulated heat wave exposure, approximately 10 min each
  FEV1 will be assessed via spirometry
Forced vital capacity (FVC) | Prior to, during, and after each simulated heat wave exposure, approximately 10 min each
  FVC will be assessed via spirometry
FEV1/FVC ratio | Prior to, during, and after each simulated heat wave exposure, approximately 10 min each
  The ratio of forced expiratory volume and forced vital capacity will be assessed via spirometry

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Health Presbyterian Hospital Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes